CLINICAL TRIAL: NCT01474291
Title: Evaluation of Factors Influencing Use of RoActemra® as Monotherapy in Rheumatoid Arthritis Patients in a Real Life Setting - ACT SOLO
Brief Title: An Observational Study of RoActemra/Actemra (Tocilizumab) As Monotherapy in Rheumatoid Arthritis Patients in Routine Clinical Practice
Acronym: ACT SOLO
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27873
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Tocilizumab: Tocilizumab administered as monotherapy or in combination with other standard of care therapy according to prescribing information and normal clinical practice.
  Interventions: Biological: Tocilizumab

INTERVENTIONS:
Biological: Tocilizumab — Tocilizumab administered according to prescribing information and normal clinical practice.
  Other Names: RoActemra®; Actemra®

SUMMARY:
This prospective, multi-center, observational study will evaluate factors influencing the use of tocilizumab (RoActemra/Actemra) as monotherapy in rheumatoid arthritis patients in real life setting. Data will be collected from participants for 12 months following initiation of tocilizumab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Patients with rheumatoid arthritis for whom the rheumatologist decides to start tocilizumab in combination with DMARD or as monotherapy

Exclusion Criteria:

* Current participation in a clinical trial in rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate to severe rheumatoid arthritis participants treated with tocilizumab in routine clinical practice
Sampling Method: Probability Sample
Enrollment: 608 (Actual)
Dates: Start 2012-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (104):
- France (104):
  - Aix-les-Bains
  - Amiens
  - Angers
  - Auch
  - Aulnay-sous-Bois
  - Avignon
  - Bastia
  - Bayonne
  - Beauvais
  - Belfort
  - Belley
  - Berck
  - Besançon
  - Bobigny
  - Bois-Guillaume
  - Bondy
  - Bonneville
  - Bordeaux
  - Boulogne-Billancourt
  - Bressuire
  - Brest
  - Bry-sur-Marne
  - Caen
  - Cahors
  - Cannes
  - Carcassonne
  - Chambray-lès-Tours
  - Châteauroux
  - Clermont-Ferrand
  - Colmar
  - Compiègne
  - Corbeil-essones
  - Corbeil-Essonnes
  - Créteil
  - Denain
  - Digne-les-Bains
  - Dijon
  - Dole
  - Draguignan
  - Druex
  - Échirolles
  - Épernay
  - Évian-les-Bains
  - Évreux
  - Évry
  - Freyming-Merlebach
  - Fréjus
  - Gap
  - Gleizé
  - Haguenau
  - Ivry-sur-Seine
  - Laon
  - Lavaur
  - Le Bouscat
  - Le Coudray
  - Le Kremlin-Bicêtre
  - Libourne
  - Liévin
  - Lille
  - Limoges
  - Lomme
  - Lyon
  - Maisons-Laffitte
  - Marseille
  - Metz-Tessy
  - Montauban
  - Montpellier
  - Moulins
  - Mulhouse
  - Nanterre
  - Nantes
  - Narbonne
  - Nevers
  - Nice
  - Nîmes
  - Orange
  - Paris
  - Perpignan
  - Périgueux
  - Pierre-Bénite
  - Poissy
  - Pontoise
  - Reims
  - Rennes
  - Rodez
  - Roubaix
  - Saint-Brieuc
  - Saint-Chamond
  - Saint-Mandé
  - Saint-Priest-en-Jarez
  - Salon-de-Provence
  - Ste Maxime
  - Strasbourg
  - Suresnes
  - Thionville
  - Toulon
  - Toulouse
  - Tourcoing
  - Valenciennes
  - Vandœuvre-lès-Nancy
  - Vannes
  - Villeneuve-Saint-Georges
  - Villeurbanne
  - Vlleneuve Sur Lot

REFERENCES:
- [Derived] Flipo RM, Maillefert JF, Chazerain P, Idier I, Coudert M, Tebib J. Factors influencing the use of tocilizumab as monotherapy in patients with rheumatoid arthritis in a real-life setting: results at 1 year of the ACT-SOLO study. RMD Open. 2017 Jan 10;3(1):e000340. doi: 10.1136/rmdopen-2016-000340. eCollection 2017. PMID 28123778

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were not allocated to study arms but were separated according to therapy regimen post hoc for efficacy and safety analyses. Of the 608 participants enrolled 5 were not eligible for analysis (1 was found to be duplicate and 4 did not receive tocilizumab infusion).
Groups:
- All Tocilizumab: Tocilizumab (RoActemra/Actemra) administered as monotherapy or in combination with other standard of care therapy according to prescribing information and normal clinical practice.
Period: Overall Study
Arm/Group | All Tocilizumab
Started | 603
Evaluable for Efficacy | 577 (Received tocilizumab infusion and met all inclusion/exclusion criteria)
Completed | 383
Not Completed | 220
Not completed — Not Evaluable for Efficacy | 26
Not completed — Lack of Treatment Efficacy | 88
Not completed — Adverse Event | 53
Not completed — Lost to Follow-up | 29
Not completed — Patient No Longer Wanted to Participate | 12
Not completed — No Reason Reported | 10
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: Efficacy population, defined as all participants who received at least one infusion of tocilizumab and who met all inclusion and exclusion criteria.
Groups:
- Tocilizumab Monotherapy: Tocilizumab administered as monotherapy according to prescribing information and normal clinical practice.
- Tocilizumab Combination Therapy: Tocilizumab administered in combination with other standard of care therapy according to prescribing information and normal clinical practice.
- Total: Total of all reporting groups
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy | Total
Number analyzed (Participants) | 228 | 349 | 577
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (12.7) | 55.3 (12.5) | 56.8 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 274 | 454
  Male | 48 | 75 | 123

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Assigned Tocilizumab Monotherapy Versus Tocilizumab as Part of Combination Therapy at Study Inclusion
Description: The number of participants assigned to tocilizumab monotherapy versus tocilizumab combination therapy is reported. A multivariate analysis was performed to search for predictive factors for the initiation of tocilizumab in monotherapy.
Time Frame: Day 1
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- All Tocilizumab: Tocilizumab administered as monotherapy or in combination with other standard of care therapy according to prescribing information and normal clinical practice.
Arm/Group | All Tocilizumab
Number analyzed (Participants) | 577
participants
  Monotherapy | 228
  Combination Therapy | 349
Statistical Analysis 1: Comparison: All Tocilizumab; Influence of baseline factor "Patient's Age (>=65)" upon physician's decision to initiate tocilizumab monotherapy (multivariate analysis); Test type: Superiority or Other; p = 0.0230, Wald Chi-square; Wald Chi-square Test for Type 3 generalized estimating equation (GEE) Analysis; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.06 to 2.30]
Statistical Analysis 2: Comparison: All Tocilizumab; Influence of baseline factor "No methotrexate (MTX) sequences within the two last years" upon physician's decision to initiate tocilizumab monotherapy (multivariate analysis); Test type: Superiority or Other; p < 0.0001, Wald Chi-square; Wald Chi-square Test for Type 3 GEE Analysis; Odds Ratio (OR) = 5.74, 95% CI 2-sided [3.92 to 8.43]
Statistical Analysis 3: Comparison: All Tocilizumab; Influence of baseline factor "Past history of severe infectious disease" upon physician's decision to initiate tocilizumab monotherapy (multivariate analysis); Test type: Superiority or Other; p = 0.0212, Wald Chi-square; Wald Chi-square Test for Type 3 GEE Analysis; Odds Ratio (OR) = 2.03, 95% CI 2-sided [1.11 to 3.70]
Statistical Analysis 4: Comparison: All Tocilizumab; Influence of baseline factor "Higher Disease Activity Score Based on 28-joint Count and Erythrocyte Sedimentation Rate (DAS28-ESR) (unit=1)" on physician decision to initiate tocilizumab monotherapy; DAS28-ESR was calculated from the number of swollen joints and tender joints using 28-joint count, ESR (millimeters per hour [mm/hour]) and patient's global assessment of disease activity; scores range from 0 to 10; higher scores correspond to greater disease activity (multivariate analysis); Test type: Superiority or Other; p = 0.0076, Wald Chi-square; Wald Chi-square Test for Type 3 GEE Analysis; Odds Ratio (OR) = 1.22, 95% CI 2-sided [1.05 to 1.41]

2. Secondary Outcome: Percentage of Participants Receiving Tocilizumab Monotherapy Who Discontinued Methotrexate (MTX)
Description: The percentage of participants who discontinued MTX treatment prior to being assigned to tocilizumab monotherapy is presented by reason for discontinuation.
  Reason for discontinuation "Other Intolerance" = intolerance other than cytopenia or hepatic cytolysis.
Time Frame: Day 1 (assessment of discontinuations within prior 2 years)
Population: Participants in the Tocilizumab Monotherapy group (Efficacy population) who discontinued MTX and with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy
Number analyzed (Participants) | 206
percentage of participants
  Therapeutic escape | 12.6
  Cytopenia | 4.4
  Hepatic Cytolysis | 20.4
  Other Intolerance | 46.1
  Patient's Choice | 4.9
  Primary Failure | 8.7
  Remission | 0.5
  Reason Not Specified | 2.4

3. Secondary Outcome: Percentage of Participants Receiving Tocilizumab Monotherapy Who Discontinued Leflunomide
Description: The percentage of participants who discontinued leflunomide treatment prior to being assigned to tocilizumab monotherapy is presented by reason for discontinuation.
Time Frame: Day 1 (assessment of discontinuations within prior 2 years)
Population: Participants in the Tocilizumab Monotherapy group (Efficacy population) who discontinued leflunomide and with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy
Number analyzed (Participants) | 34
percentage of participants
  Therapeutic escape | 17.6
  Intolerance | 47.1
  Patient's Choice | 2.9
  Primary Failure | 32.4

4. Secondary Outcome: Percentage of Participants Receiving Tocilizumab Monotherapy Who Discontinued Sulfasalazine
Description: The percentage of participants who discontinued sulfasalazine treatment prior to being assigned to tocilizumab monotherapy is presented by reason for discontinuation.
Time Frame: Day 1 (assessment of discontinuations within prior 2 years)
Population: Participants in the Tocilizumab Monotherapy group (Efficacy population) who discontinued sulfasalazine and with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy
Number analyzed (Participants) | 17
percentage of participants
  Therapeutic escape | 23.5
  Intolerance | 41.2
  Primary failure | 35.3

5. Secondary Outcome: Percentage of Participants Receiving Tocilizumab Monotherapy Who Discontinued Hydroxychloroquine
Description: The percentage of participants who discontinued hydroxychloroquine treatment prior to being assigned to tocilizumab monotherapy is presented by reason for discontinuation.
Time Frame: Day 1 (assessment of discontinuations within prior 2 years)
Population: Participants in the Tocilizumab Monotherapy group (Efficacy population) who discontinued hydroxychloroquine and with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy
Number analyzed (Participants) | 10
percentage of participants
  Therapeutic escape | 30.0
  Primary failure | 50.0
  Reason Not Specified | 20.0

6. Secondary Outcome: Percentage of Participants Receiving Tocilizumab Monotherapy Who Discontinued Unspecified Conventional Synthetic Disease-modifying Antirheumatic Drugs (csDMARDs)
Description: The percentage of participants who discontinued treatment with unspecified csDMARDs prior to being assigned to tocilizumab monotherapy is presented by reason for discontinuation.
Time Frame: Day 1 (assessment of discontinuations within prior 2 years)
Population: Participants in the Tocilizumab Monotherapy group (Efficacy population) who discontinued treatment with unspecified csDMARDs and with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy
Number analyzed (Participants) | 79
percentage of participants
  Therapeutic escape | 26.6
  Intolerance | 38.0
  Patient's Choice | 1.3
  Primary Failure | 27.8
  Remission | 1.3
  Reason Not Specified | 5.1

7. Secondary Outcome: Mean Number of Tocilizumab Infusions Over the Study Period
Time Frame: Up to 30 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: infusions
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 228 | 349
infusions | 9.1 (4.3) | 9.7 (4.0)

8. Secondary Outcome: Percentage of Participants Who Received Tocilizumab Infusions Over the Study Period
Description: The percentage of participants who received infusions is presented by category of total infusions received over the study period.
Time Frame: Up to 13.4 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 228 | 349
percentage of participants
  1 Infusion | 5.7 | 4.6
  2 Infusions | 4.8 | 4.0
  3 Infusions | 7.0 | 2.6
  4 Infusions | 3.5 | 4.0
  5 Infusions | 4.8 | 5.7
  6 Infusions | 3.9 | 5.4
  7 Infusions | 6.6 | 2.6
  8 Infusions | 3.5 | 2.6
  9 Infusions | 2.6 | 5.4
  10 Infusions | 4.4 | 5.4
  11 Infusions | 7.9 | 6.3
  12 Infusions | 16.7 | 22.3
  13 Infusions | 17.1 | 18.3
  14 Infusions | 11.0 | 9.7
  15 Infusions | 0.4 | 0.9

9. Secondary Outcome: Percentage of Participants With No Modification of Tocilizumab Treatment Over the Study Period
Description: The percentage of participants with no modifications (dose modification or discontinuation) is presented.
Time Frame: Up to 30 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 228 | 349
percentage of participants | 48.2 | 56.2

10. Secondary Outcome: Percentage of Participants With at Least One csDMARD Intensification During the Study
Description: csDMARD intensification was defined as an addition of a csDMARD without suppression of other csDMARD, dose increase of a csDMARD, switch (addition and suppression) of a csDMARD without intolerance, biological abnormality or symptom improvement to the suppressed csDMARD, or modification of the MTX administration route (from oral route to intramuscular/subcutaneous) with dose increase or maintenance.
Time Frame: Up to 30 months
Population: Participants in Efficacy population who received at least 1 infusion of tocilizumab, who met all inclusion/exclusion criteria, and with no permanent discontinuation of tocilizumab treatment over the study period. For efficacy criteria with response/non response values, participants with non-evaluable response were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 158 | 256
percentage of participants | 8.2 | 4.7

11. Secondary Outcome: Percentage of Participants in Disease Activity Score Based on 28-joint Count and Erythrocyte Sedimentation Rate (DAS28-ESR) Low Disease Activity (LDA) at Month 12
Description: DAS28-ESR was calculated from the number of swollen joints and tender joints using the 28-joint count, ESR (mm/hour) and patient's global assessment of disease activity; scores range from 0 to 10, where lower scores indicate less disease activity. A score of ≤3.2 was considered to be DAS28-ESR LDA. Participants with missing data were considered to have failed to achieve the outcome.
Time Frame: Month 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 228 | 349
percentage of participants | 41.2 | 44.4

12. Secondary Outcome: Percentage of Participants With DAS28-ESR Remission at Month 12
Description: DAS28-ESR was calculated from the number of swollen joints and tender joints using the 28-joint count, ESR (mm/hour) and patient's global assessment of disease activity; scores range from 0 to 10, where lower scores indicate less disease activity. A score of <2.6 was considered to be DAS28-ESR remission. Participants with missing data were considered to have failed to achieve the outcome.
Time Frame: Month 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 228 | 349
percentage of participants | 34.6 | 35.5

13. Secondary Outcome: Percentage of Participants With Clinical Disease Activity Index (CDAI) LDA at Month 12
Description: CDAI was calculated from the number of swollen joints and tender joints using the 28-joint count and the patient's global assessment of disease activity and physician's global assessment of disease activity; CDAI scores range from 0 to 76, where lower scores indicate less disease activity. A score of ≤10 was considered to be CDAI LDA. Participants with missing data were considered to have failed to achieve the outcome.
Time Frame: Month 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 228 | 349
percentage of participants | 31.1 | 23.5

14. Secondary Outcome: Percentage of Participants With CDAI Remission at Month 12
Description: CDAI was calculated from the number of swollen joints and tender joints using the 28-joint count and the patient's global assessment of disease activity and physician's global assessment of disease activity; CDAI scores range from 0 to 76, where lower scores indicate less disease activity. A score of ≤2.8 was considered to be CDAI remission. Participants with missing data were considered to have failed to achieve the outcome.
Time Frame: Month 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 228 | 349
percentage of participants | 9.6 | 8.6

15. Secondary Outcome: Percentage of Participants With Simplified Disease Activity Index (SDAI) LDA at Month 12
Description: SDAI was calculated from the number of swollen joints and tender joints using the 28-joint count, C-reactive protein (CRP) (milligrams per liter (mg/L)) per , and the patient's global assessment of disease activity and physician's global assessment of disease activity; SDAI scores range from 0 to 86, where lower scores indicate less disease activity. A score of ≤11 was considered to be SDAI LDA. Participants with missing data were considered to have failed to achieve the outcome.
Time Frame: Month 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 228 | 349
percentage of participants | 30.7 | 23.2

16. Secondary Outcome: Percentage of Participants With SDAI Remission at Month 12
Description: SDAI was calculated from the number of swollen joints and tender joints using the 28-joint count, CRP (mg/L), and the patient's global assessment of disease activity and physician's global assessment of disease activity; SDAI scores range from 0 to 86, where lower scores indicate less disease activity. A score of ≤3.3 was considered to be SDAI remission. Participants with missing data were considered to have failed to achieve the outcome.
Time Frame: Month 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 228 | 349
percentage of participants | 10.1 | 9.7

17. Secondary Outcome: Percentage of Participants With American College or Rheumatology (ACR)20, ACR50, and ACR70 at Month 12
Description: ACR20/50/70 response was calculated as improvement (from baseline) of at least 20/50/70% (respectively) of tender and of swollen joints, and improvement from baseline of least 20/50/70% (respectively) in at least 3 of the 5 following parameters: participant's pain assessment, patient's global assessment of disease activity, physician's global assessment of disease activity, health assessment questionnaire disability index (HAQ-DI) score, and ESR (mm/hour) or CRP (mg/L). Participants with missing data were considered to have failed to achieve the outcome.
Time Frame: Month 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 228 | 349
percentage of participants
  ACR20 | 32.5 | 26.4
  ACR50 | 21.9 | 16.9
  ACR70 | 9.6 | 9.7

18. Secondary Outcome: Percentage of Participants With Good or Moderate European League Against Rheumatism (EULAR) Response at Month 12
Description: EULAR response was categorized as good or moderate response and was calculated as the difference between DAS28-ESR scores at baseline and Month 12. DAS28-ESR was calculated from the number of swollen joints and tender joints using the 28-joint count, ESR (mm/hour) and patient's global assessment of disease activity; scores range from 0 to 10, where lower scores indicate less disease activity.
  * If diminution from baseline >1.2 and score ≤3.2 at Month 12 = good response
  * If diminution from baseline >1.2 and score >3.2 at Month 12 = moderate response
  * If diminution from baseline >0.6 and ≤1.2, and score ≤5.1 at Month 12 = moderate response
  * If diminution from baseline >0.6 and ≤1.2, and score >5.1 at Month 12 = non-response
  * If diminution from baseline ≤1.2 at Month 12 = non-response
  * Participants with missing data were considered as non-response
Time Frame: Month 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 228 | 349
percentage of participants
  Good Response | 40.4 | 38.7
  Moderate Response | 9.6 | 10.9

19. Secondary Outcome: Mean Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score
Description: The HAQ-DI is a participant-reported assessment of ability to perform daily living activities. This composite index score ranges from 0 (normal) to 3 (total functional disability) and includes questions regarding 8 domains (dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week). A decrease in score corresponds to improvement in participant-assessed health state.
Time Frame: Baseline; Month 6; Month 12
Population: Participants in the Efficacy population who received at least one infusion of tocilizumab, who met all inclusion and exclusion criteria, and with available data at the respective time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 228 | 349
units on a scale
  Baseline (n = 171, 251) | 1.62 (0.67) | 1.47 (0.66)
  Change at Month 6 (n = 85, 121) | -0.45 (0.64) | -0.44 (0.62)
  Change at Month 12 (n = 74, 106) | -0.47 (0.68) | -0.45 (0.62)

20. Secondary Outcome: Mean Change From Baseline in Rheumatoid Arthritis Impact of Disease (RAID) Score
Description: The RAID questionnaire is a participant-reported outcome measure evaluating the impact of rheumatoid arthritis on participant quality of life. This composite index score ranges from 0 (best) to 10 (worst) and includes questions regarding 7 domains (pain, functional disability assessment, fatigue, sleep, physical well-being, emotional well-being, coping). A decrease in score corresponds to improvement in participant-assessed health state.
Time Frame: Baseline; Month 6, Month 12
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 228 | 349
units on a scale
  Baseline (n = 170, 252) | 6.47 (1.98) | 5.92 (1.89)
  Change at Month 6 (n = 82, 122) | -2.11 (2.23) | -2.07 (2.47)
  Change at Month 12 (n = 72, 108) | -2.42 (2.29) | -2.15 (2.34)

21. Secondary Outcome: Percentage of Participants With Acceptable Health State Assessed by the Patient Acceptable Symptom State (PASS) Questionnaire.
Description: Participants were asked: "If you were to remain in the same condition for the next few months as you have been over the last 8 days, would this be 1) acceptable, 2) unacceptable?" The percentage of participants who responded "acceptable" at each time point is presented.
Time Frame: Baseline; Month 6; Month 12
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 228 | 349
percentage of participants
  Baseline (n = 168, 246) | 25.6 | 34.1
  Month 6 (n = 101, 153) | 69.3 | 73.2
  Month 12 (n = 84, 132) | 84.5 | 79.5

22. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event was defined as any unfavorable and unintended sign (including an abnormal laboratory finding if accompanied by clinical symptoms, results in a change in study treatment, results in a medical intervention or a change in concomitant therapy or clinically significant in the investigator's judgment), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Up to 30 months
Population: Safety population, defined as participants who received at least one infusion of tocilizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Number analyzed (Participants) | 234 | 369
percentage of participants | 54.7 | 53.4

ADVERSE EVENTS:
Time Frame: Up to 30 months
Description: Safety population, defined as participants who received at least one infusion of tocilizumab.
Arm/Group | Tocilizumab Monotherapy | Tocilizumab Combination Therapy
Serious Adverse Events (participants affected / at risk) | 31/234 | 43/369
Other Adverse Events (participants affected / at risk) | 112/234 | 182/369
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Monotherapy (N=234) | Tocilizumab Combination Therapy (N=369)
Bronchitis (Infections and infestations) | 0 | 4
Device related infection (Infections and infestations) | 1 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 2
Anal abscess (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Bursitis infective staphylococcal (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Ecthyma (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Infected varicose vein (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic arthritis staphylococcal (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tongue abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Viral rash (Infections and infestations) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Sigmoiditis (Gastrointestinal disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Coronary artery thrombosis (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Demyelination (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Sciatic nerve palsy (Nervous system disorders) | 0 | 1
Device dislocation (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Inflammation (General disorders) | 1 | 0
Medical device pain (General disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Keratolysis exfoliative acquired (Skin and subcutaneous tissue disorders) | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 1
Osteosynthesis (Surgical and medical procedures) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Acquired haemophilia (Blood and lymphatic system disorders) | 0 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Fallopian tube cyst (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Monotherapy (N=234) | Tocilizumab Combination Therapy (N=369)
Bronchitis (Infections and infestations) | 18 | 23
Nasopharyngitis (Infections and infestations) | 7 | 9
Tonsillitis (Infections and infestations) | 6 | 6
Urinary tract infection (Infections and infestations) | 6 | 5
Oral herpes (Infections and infestations) | 5 | 4
Sinusitis (Infections and infestations) | 6 | 3
Gastroenteritis (Infections and infestations) | 1 | 7
Paronychia (Infections and infestations) | 4 | 4
Influenza (Infections and infestations) | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 4
Lung infection (Infections and infestations) | 1 | 4
Pharyngitis (Infections and infestations) | 1 | 4
Erysipelas (Infections and infestations) | 2 | 2
Pneumonia (Infections and infestations) | 0 | 4
Rhinitis (Infections and infestations) | 2 | 2
Escherichia urinary tract infection (Infections and infestations) | 2 | 1
Furuncle (Infections and infestations) | 1 | 2
Gastroenteritis viral (Infections and infestations) | 2 | 1
Oral fungal infection (Infections and infestations) | 1 | 2
Tooth infection (Infections and infestations) | 2 | 1
Bronchopneumonia (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 2 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 2
Ear infection (Infections and infestations) | 1 | 1
Herpes virus infection (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 1 | 1
Infected bites (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 0 | 2
Tinea pedis (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 1
Acarodermatitis (Infections and infestations) | 0 | 1
Bacterial prostatitis (Infections and infestations) | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 1
Bursitis infective (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Eyelid infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1
Genital herpes (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 0 | 1
Infected dermal cyst (Infections and infestations) | 1 | 1
Laryngitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 0 | 1
Onychomycosis (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 1
Prostatitis Escherichia coli (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 1
Sinobronchitis (Infections and infestations) | 1 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Superinfection (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0
Viral rhinitis (Infections and infestations) | 1 | 0
Viral tonsillitis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 25 | 31
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 4
Leukopenia (Blood and lymphatic system disorders) | 1 | 3
Blood disorder (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Asthenia (General disorders) | 3 | 15
Fatigue (General disorders) | 2 | 2
Pyrexia (General disorders) | 2 | 2
Chest pain (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 1 | 2
Adverse event (General disorders) | 0 | 2
Chest discomfort (General disorders) | 1 | 1
Feeling hot (General disorders) | 1 | 1
Drug ineffective (General disorders) | 0 | 1
Drug intolerance (General disorders) | 1 | 0
Face oedema (General disorders) | 0 | 1
Facial pain (General disorders) | 1 | 0
Haemorrhagic cyst (General disorders) | 1 | 0
Hot flush (General disorders) | 0 | 1
Hyperthermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Infusion site pain (General disorders) | 0 | 1
Infusion site warmth (General disorders) | 1 | 0
Local swelling (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Nodule (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Papillitis (General disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 9
Diarrhoea (Gastrointestinal disorders) | 2 | 8
Nausea (Gastrointestinal disorders) | 6 | 4
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 9
Abdominal pain upper (Gastrointestinal disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 0 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 4
Eczema (Skin and subcutaneous tissue disorders) | 3 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rebound psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone erosion (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint adhesion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Weight increased (Investigations) | 6 | 2
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Transaminases increased (Investigations) | 1 | 1
Biopsy skin (Investigations) | 0 | 1
Blood pressure decreased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Colonoscopy (Investigations) | 0 | 1
Creatinine renal clearance increased (Investigations) | 1 | 0
Eosinophil count increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Laboratory test abnormal (Investigations) | 1 | 0
Lipids abnormal (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Low density lipoprotein increased (Investigations) | 1 | 0
Neutrophil count increased (Investigations) | 0 | 1
Red blood cells urine positive (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 8 | 11
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 1
Headache (Nervous system disorders) | 5 | 7
Sciatica (Nervous system disorders) | 2 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1
Foot operation (Surgical and medical procedures) | 0 | 3
Tooth extraction (Surgical and medical procedures) | 2 | 1
Cataract operation (Surgical and medical procedures) | 1 | 1
Blepharoplasty (Surgical and medical procedures) | 1 | 0
Bunion operation (Surgical and medical procedures) | 1 | 0
Colon polypectomy (Surgical and medical procedures) | 0 | 1
Cyst removal (Surgical and medical procedures) | 0 | 1
Dental care (Surgical and medical procedures) | 0 | 1
Dental implantation (Surgical and medical procedures) | 0 | 1
Drug therapy changed (Surgical and medical procedures) | 1 | 0
Elbow operation (Surgical and medical procedures) | 0 | 1
Gingival graft (Surgical and medical procedures) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Lymphadenectomy (Surgical and medical procedures) | 1 | 0
Salivary gland calculus removal (Surgical and medical procedures) | 1 | 0
Skin neoplasm excision (Surgical and medical procedures) | 1 | 0
Tonsillectomy (Surgical and medical procedures) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 4
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Skin wound (Injury, poisoning and procedural complications) | 1 | 1
Wound (Injury, poisoning and procedural complications) | 2 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 1
Drug dose omission (Injury, poisoning and procedural complications) | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0
Eyelid injury (Injury, poisoning and procedural complications) | 1 | 0
Foetal exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 2
Haematoma (Vascular disorders) | 1 | 1
Procedural hypertension (Vascular disorders) | 2 | 0
Flushing (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Phlebitis superficial (Vascular disorders) | 1 | 0
Varicose ulceration (Vascular disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 2 | 2
Uveitis (Eye disorders) | 1 | 1
Vision blurred (Eye disorders) | 0 | 2
Dry eye (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 5 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 2
Palpitations (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 4
Depression (Psychiatric disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 2
Allergy to vaccine (Immune system disorders) | 0 | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Social problem (Social circumstances) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.